CLINICAL TRIAL: NCT00967486
Title: Selective Shunting in Appropriately Selected Patients Undergoing Carotid Endarterectomy Based on Stump Pressure
Brief Title: Selective Versus Routine Shunting in Carotid Endarterectomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Ali AbuRahma, Ali Fawzi AbuRahma MD, Vascular Center of Excellence(CAMC Medical Staff - with admitting privileges)., CAMC Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-11-1878
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Results first posted 2013-10-24 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-08

CONDITIONS: Stenoses, Carotid Artery
MeSH Terms: conditions — Carotid Stenosis | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine Shunt (Active Comparator): These patients are called routine as the routine method of carotid endarterectomy is used.
  Interventions: Procedure: Carotid endarterectomy with routine shount
- Selective Shunt (Active Comparator): These patients are selectively used for shunting or not shunting based on systolic pressure < 40mmHg. This group is further used as subgroup analysis.
  Interventions: Procedure: Carotid endarterectomy with selective shunt

INTERVENTIONS:
Procedure: Carotid endarterectomy with routine shount
  Arms: Routine Shunt
Procedure: Carotid endarterectomy with selective shunt
  Arms: Selective Shunt

SUMMARY:
The project involves prospectively randomizing patients to either routine carotid shunting or selective carotid shunting during Carotid endarterectomy (CEA) under general anesthesia (GA) to see the difference in post-op complications and occurence rates. Patients will be randomized to Routine shunt vs selective groups.

DETAILED DESCRIPTION:
The significance extends to all surgeons who perform Carotid endarterectomy because of their desire to improve patient care by decreasing the overall perioperative complication rate of the procedure by selectively not shunting those patients who ideally do not require it and thus eliminating the attendant morbidity associated with it.

The hypothesis is that there will be no difference in patient outcomes (death, minor strokes, major strokes, transient ischemic attack (TIA)) for patients undergoing a Carotid endarterectomy with a SP of > 50 mm Hg using selective shunting.Patients will be randomized to Routine shunt vs selective groups. In Selective shunt, there will be subgroup analysis to measure % stenosis if the systolic pressure is < 40mmHg calling it as Shunt group. All patients in the study, irrespective of treatment group will be followed post-operatively from 24 hours to 30 days. The patient will be monitored and the following outcomes documented - death, minor stroke, major stroke, trans-ischemic attack (TIA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a SP >= 50 mmHg will be randomized to receive a shunt or not receive a shunt.

Exclusion Criteria:

* Patients that will be excluded are those who present for a redo CEA, have had a coronary artery bypass graft (CABG), permanent stroke, and or a contralateral artery total occlusion of > 30%.
* Finally, consented patients with a stump pressure of <= 50 mm Hg will be excluded from the study and receive standard of care.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali F AbuRhama, M.D., Principal Investigator — CAMC Medical Staff - with admitting privileges
Locations (1):
- (Vascular Center of Excellence), Charleston, West Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Routine Shunt: Routine method of CEA
- Selective Shunt: Selective method if CEA with based Systolic pressure 40 mmHg
Period: Overall Study
Arm/Group | Routine Shunt | Selective Shunt
Started | 98 | 102
Completed | 98 | 102
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Routine Shunt: routine methods of CEA
- Total: Total of all reporting groups
Arm/Group | Routine Shunt | Selective Shunt | Total
Number analyzed (Participants) | 98 | 102 | 200
Age, Categorical [Count of Participants; unit: Participants]
  Between 18 and 65 years | 38 | 44 | 82
  >=65 years | 60 | 58 | 118
Age Continuous [Mean (Standard Deviation); unit: years] | 68.78 (9.08) | 67.29 (9.81) | 68.02 (9.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 53 | 103
  Male | 48 | 49 | 97
Region of Enrollment [Number; unit: participants]
  United States | 98 | 102 | 200

OUTCOME MEASURES:

1. Primary Outcome: Overall Perioperative Complications Between Selective vs. Routine Shunting.
Description: perioperative complication included at least one of transient ischemic attack (TIA), hemorrhage, myocardial infarction [MI], or asymptomatic carotid thrombosis or congestive heart failure.
Time Frame: Within 30 days of enrollment
Measure: Number; unit: Participants
Arm/Group | Routine Shunt | Selective Shunt
Number analyzed (Participants) | 98 | 102
Participants | 7 | 8
Statistical Analysis 1: Comparison: Routine Shunt vs Selective Shunt; Test type: Superiority or Other; p < 0.05, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Routine Shunt | Selective Shunt
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No